CLINICAL TRIAL: NCT04360291
Title: Impact de la Restriction du Champ Visuel Sur l'Exploration Visuelle
Brief Title: Impact of Visual Field Restriction on Visual Exploration
Acronym: REVE
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Centre Hospitalier National d'Ophtalmologie des Quinze-Vingts (Other)
Responsible Party: Sponsor
Other Study IDs: P19-05; 2019-A01198-49 (Other: N°IDRCB)
Record Dates: First submitted 2019-10-23; First posted 2020-04-24 (Actual); Last update posted 2020-04-24 (Actual); Status verified 2020-04

CONDITIONS: Pigmentary Retinopathy
MeSH Terms: conditions — Retinitis Pigmentosa

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Healthy volunteers: Healthy volunteers
  Interventions: Other: Eye tracker
- Retinopathy pigment: Patients with retinopathy pigment
  Interventions: Other: Eye tracker

INTERVENTIONS:
Other: Eye tracker — In visual search tasks, participants will sit in front of a screen and observe during each visual scene for a maximum of 45 seconds. Their eye movements will be recorded

SUMMARY:
To communicate with the observer and guide his gaze on the canvas, painters have developed different stylistic processes that artists, in the manner of scientists, have acquired on the functioning of human visual perception. This direct communication between the artist and the observer is strongly impacted for people with visual impairments.

In order to improve the accessibility and autonomy of visually impaired people in museums and to allow each observer to feel the visual and emotional experience closest to the original work of the artist, it is essential to identify the modifications. perceptive generated by the constriction of vision

DETAILED DESCRIPTION:
In this experiment, the investigators study the adaptive strategies developed by people with retinitis pigmentosa in the perception of figurative works of art. Peripheral vision is crucial for detecting objects and directing attention to the relevant areas of the environment, while central vision, of high spatial resolution, is especially essential for identifying the nature of objects. The integration of perceived information in peripheral vision and central vision makes it possible to quickly and effortlessly develop a spatial representation of the environment, to activate categorical knowledge on the observed scene and to relate the various objects perceived. However, with the progressive constriction of the visual field, the visual exploration of the subject RP can not be carried out with the strategies used by the healthy subjects, in which the targets of the saccades are in particular determined according to the information perceived in peripheral vision.

Through the recording of eye movements, the investigators compare the differences in visual explorations of people with retinitis pigmentosa and healthy people with or without a simulated deficit.

ELIGIBILITY:
Groupe 1

Inclusion Criteria:

* no visual pathology
* Age ≥ 18 and <65 years
* Binocular visual acuity ≥8 / 10th or ≤ +0.10 logMAR
* Comprehension of the written and spoken French language
* Signed consent to participate in the study
* Health insurance affiliation
* Visit to an ophthalmologist less than a year old

Exclusion Criteria:

* Pregnant or lactating woman
* Ocular pathology that may interfere with planned assessments
* Treatment that may interfere with planned assessments
* Participation in another study that may interfere with this study.
* Severe pathology unbalanced or interfering with planned assessments.
* Neurological deficit including history of epileptic pathology, photosensitive epilepsy, sensory-motor coordination disorders, vestibular or cerebellar pathology
* Inability to give consent personally.
* Adults protected by law.

Groupe 2

Inclusion Criteria:

* Retinopathy pigmentary dystrophy rods-cones.
* Binocular visual acuity ≥4 / 10 (≤0.4 logMAR).
* Horizontal diameter of the residual Goldmann field of view ≤ 25 ° of binocular diameter at III4.
* Comprehension of the French language, written or oral.
* Signed consent
* Visual assessment less than 6 months old

Exclusion Criteria:

* Pregnant or nursing woman.
* Ocular pathology that may interfere with planned assessments.
* Treatment that may interfere with planned assessments.
* Severe pathology unbalanced or interfering with planned assessments.
* Participation in another study that may interfere with this study.
* Neurological deficit including antecedent of epileptic pathology, photosensitive epilepsies, non-visual sensory disturbances, motor disorders, or sensorimotor coordination disorders, vestibular or cerebellar pathology.
* Inability to give consent personally.
* Adults protected by law.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Subjects with pigmentary retinopathy
Sampling Method: Non-Probability Sample
Enrollment: 45 (Estimated)
Dates: Start 2019-11-04 (Actual); Primary Completion 2020-09-11 (Estimated); Study Completion 2021-10-17 (Estimated)

PRIMARY OUTCOMES:
Eye movements | through study completion,, an average of 1 year
  Eye movements will be recorded by an eye trackervisual impairment whose peripheral visual field is masked
  They will be invited to observe scenes of human interaction presented on photographs, pictorial works or artificial scenes with or without prior instruction.
  In addition to the elementary variables recorded during the exploration by these subjects, such as the number, the amplitude or the orientation of the saccades, the sequence of fixations will be analyzed to define the exploratory strategy used.
Fixation strategy | through study completion,, an average of 1 year
  The fixation strategy characterized by the path of the gaze of the subjects on the screen to locate the targets.
Target location accuracy | through study completion,, an average of 1 year
  Target location accuracy, defined by the distance between the point of re-fixation on the target and the actual position of the target

CONTACTS AND LOCATIONS:
Overall Officials: Avinoam Safran, Principal Investigator — Institut de la vision
Locations (1):
- Institut de la vision, Paris, France